CLINICAL TRIAL: NCT04663412
Title: Indocyanine Green Fluorescence Imaging, Sentinel Lymph Node Mapping in Patients With Vulvar Cancer: Peritumoral Injection Dosage and Waiting Times in Our Experience
Brief Title: Indocyanine Green Fluorescence Imaging, Sentinel Lymph Node Mapping in Patients With Vulvar Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera per l'Emergenza Canizzaro (Other)
Responsible Party: Principal Investigator, Paolo Scollo, Professor, Azienda Ospedaliera per l'Emergenza Canizzaro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8337
Record Dates: First submitted 2020-12-01; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Vulvar Cancer
Keywords: vulvar cancer; indocyanine green; sentinel node; surgery; single center
MeSH Terms: conditions — Vulvar Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients FIGO IB stage (Experimental): Vulvar Cancer IB stage
  Interventions: Other: Sentinel lymph node mapping with indocyanine green fluorescence imaging in vulvar cancer (FIGO Stage IB)

INTERVENTIONS:
Other: Sentinel lymph node mapping with indocyanine green fluorescence imaging in vulvar cancer (FIGO Stage IB) — Patients diagnosed with vulvar squamous cell carcinoma (FIGO IB stage) underwent bilateral radical vulvectomy, SLN search and removal, and bilateral inguinal lymphadenectomy at the Cannizzaro Hospital Operative Unit of Obstetrics and Gynecology Department (Catania, Italy). 3 ml of indocyanine green (ICG) 0.5 mg/mL was administered in 3 peritumoral injections under general anesthesia to screen the SLN. The images were acquired using an intraoperative infrared camera system, which allowed intraoperative visualization of the SLN. An SLN was identified for each patient. The lymph nodes examined by the pathologist were negative for metastatic localization of the disease. However, patients underwent bilateral inguinofemoral lymphadenectomy, as this procedure is not currently codified as a gold standard for the detection of SLN in vulvar cancer.

SUMMARY:
The potential of the administration of indocyanine green (ICG) allows the execution of SLN biopsy, avoiding the multiple administrations of radiocolloid in the pre-operative phase, painful for the patient, elimination, and exposure to radioactivity. Therefore, while requiring standardization of the methodology and a large-scale application, this procedure could open a new surgical management perspective in patients with early-stage vulvar cancer.

DETAILED DESCRIPTION:
According to The European Society of Gynaecological Oncology (ESGO) guidelines, the investigators decided to treat patients with vulvar squamous cell carcinoma (vSCC), FIGO stage IB with radical vulvectomy, sentinel lymph node search, and removal with indocyanine green (ICG) subsequent bilateral inguinofemoral lymphadenectomy.

Intraoperative imaging system The SPY Portable Handheld Imager (SPY-PHI) © Stryker was used as the intraoperative imaging device. This device uses SPY fluorescence imaging technology to visually assess blood circulation in blood vessels and associated tissue perfusion during surgery. The design of SPY-PHI makes the device versatile, enabling the operator to frame the operating field and use the acquired images in real-time, integrating fluorescence signal data with white light images in real-time. The SPY Portable Handheld Imaging System Camera, with integrated optics and cables for real-time fluorescence imaging in visible light and near-infrared, is ideal for open surgery.

Intraoperative detection of the sentinel lymph node The fluorescent agent was administered to patients placed in the lithotomy position under general anesthesia. Indocyanine green (ICG) prepared with a 25 mg vial of green indocyanine green (ICG) (Pulsion Medical Systems AG, Munich, Germany) diluted in 50 mL of water for injections (B. Braun Medical) was used, resulting in a concentration of 0.5 mg/mL. Injection of 1 ml per quadrant was administered in the three quadrants around the vulvar lesion. After the injection, the infrared camera, equipped with a movable arm, was placed in front of the patient to detect transcutaneous fluorescence during surgery. Subsequently, the SLN was localized based on the fluorescence intensity. The intraoperative fluorescence detection camera system was used to open, identify, and remove the SLN and the vulvectomy of the groin. After the excision, the capture of the residual lymphatic pathway could be seen bilaterally through the infrared camera. Additionally, all SLNs were subject to ex vivo imaging due to the presence of fluorescence. The excised SLNs were sent to pathological anatomy and processed according to the standard SLN protocol.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with vulvar squamous cell carcinoma FIGO IB stage

Exclusion Criteria:

-

Ages: 20 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2020-07-09 (Actual); Primary Completion 2021-07-20 (Estimated); Study Completion 2023-07-20 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years
  The length of time during and after the treatment of vulvar cancer with sentinel node, that a patient lives with the disease but it does not get worse.

SECONDARY OUTCOMES:
Overall Survival | 3 years
  The length of time from either the date of diagnosis or the start of treatment for vulvar cancer, that patients diagnosed with the disease are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Scollo, Prof., Principal Investigator — A.O.E. Cannizzaro
Locations (1):
- Ginecologia e Ostetricia, Catania, Italy

IPD SHARING:
Plan to Share IPD: Undecided